CLINICAL TRIAL: NCT02974257
Title: Randomized, Double-blind, Placebo-controlled Trial of the Effect of Thiamine on Oxygen Consumption After In-hospital Cardiac Arrest.
Brief Title: Thiamine vs. Placebo to Increase Oxygen Consumption After Cardiac Arrest
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study stopped early after consultation with DSMB
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Katherine Berg, Assistant Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016P000347; 1K23HL128814-01A1 (NIH)
Record Dates: First submitted 2016-11-23; First posted 2016-11-28 (Estimated); Results first posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-03

CONDITIONS: Cardiac Arrest; Shock; Lactic Acidosis; Thiamin Deficiency
Keywords: cardiac arrest; thiamine; oxygen consumption; lactate; shock
MeSH Terms: conditions — Heart Arrest; Shock; Acidosis, Lactic; Beriberi | interventions — Thiamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Thiamine (Experimental): Intervention: Thiamine 500mg IV every 12 hours for 2 days. Oxygen consumption will be monitored with a non-invasive monitor continuously for 2 days and lactate, pyruvate dehydrogenase and other routine lab values will be checked at serial time points.
  Interventions: Drug: Thiamine
- Placebo (Placebo Comparator): Intervention: Placebo (100mL normal saline) IV every 12 hours for 2 days. Oxygen consumption will be monitored with a non-invasive monitor continuously for 2 days and lactate, pyruvate dehydrogenase and other routine lab values will be checked at serial time points.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Thiamine — Thiamine 500mg IV twice daily for 2 days
  Other Names: vitamin B1
  Arms: Thiamine
Other: placebo — 100mL normal saline IV every 12 hours for 2 days
  Other Names: normal saline
  Arms: Placebo

SUMMARY:
This study is to evaluate whether thiamine can increase oxygen consumption and lower lactate in patients who initially survive an in-hospital cardiac arrest. Patients who are successfully resuscitated after an in-hospital cardiac arrest and who are on mechanical ventilation in the intensive care unit will be enrolled, and will get either thiamine or placebo. Their oxygen consumption and lactate will be measured at serial time points and compared between groups. The investigators' hypothesis is that thiamine will help restore the body's ability to metabolize oxygen normally (aerobic metabolism), leading to an increase in oxygen consumption and a decrease in lactate.

DETAILED DESCRIPTION:
In-hospital cardiac arrest often leads to shock and organ failure, and low oxygen consumption and high lactate are associated with worse outcome. Thiamine is a B vitamin necessary to maintain the body's ability to use oxygen effectively, and the investigators have found that many patients are thiamine deficient after cardiac arrest. The investigators have also found that thiamine can decrease lactate in thiamine-deficient patients who are critically ill. Patients in this study will be randomized to receive either thiamine or placebo every 12 hours for 2 days after surviving an in-hospital cardiac arrest. The investigators will measure oxygen consumption continuously during that time with a monitor attached to the ventilator tubing, and will also measure lactate and other lab values at several time points.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (age > 18 years)
* Cardiac arrest occurring while admitted to the hospital, with sustained (>20 minutes) return of spontaneous circulation (ROSC)
* Mechanically ventilated at the time of enrollment
* Within 12 hours of cardiac arrest event

Exclusion Criteria:

* Clinical indication for thiamine administration (alcoholism, known or highly suspected deficiency) or treatment with thiamine beyond the amount found in a standard multivitamin within the last 10 days
* Comfort measures only or anticipated withdrawal of support within 24 hours
* Severe agitation
* Protected populations (pregnant women, prisoners)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2022-02-07 (Actual); Study Completion 2022-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine M Berg, MD, Principal Investigator — Beth
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Thiamine | Placebo
Started | 21 | 20
Completed | 18 | 18
Not Completed | 3 | 2
Not completed — Transitioned to comfort-measures only prior to meeting fraction of inspired oxygen (FiO2) criteria | 1 | 0
Not completed — Clinical indication for thiamine | 1 | 0
Not completed — Already on thiamine | 1 | 0
Not completed — Extubated prior to study drug | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Thiamine | Placebo | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 69 [63 to 76] | 72.5 [66 to 77] | 69.5 [65 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 12 | 12 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 11 | 14 | 25
  Unknown or Not Reported | 5 | 3 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 7 | 9 | 16
  Race: Black | 3 | 4 | 7
  Race: Asian | 2 | 0 | 2
  Race: Other/Not Reported | 6 | 5 | 11
Initial Rhythm [Count of Participants; unit: Participants]
  Pulseless Electrical Activity | 13 | 12 | 25
  Asystole | 1 | 2 | 3
  Ventricular Fibrillation/Pulseless Ventricular Tachycardia | 4 | 4 | 8
Minutes to Return of Spontaneous Circulation (ROSC) [Median (Inter-Quartile Range); unit: minutes] | 11 [6 to 15] | 10.5 [6 to 15] | 11 [6 to 15]

OUTCOME MEASURES:

1. Primary Outcome: Lactate
Description: The investigators will evaluate the median lactate level over two days, compared between groups
Time Frame: 2 days
Population: A total of 5 patients in the thiamine group and 4 patients in placebo group missing lactate at 48-hours due to death; these values were imputed using a 20 percent increase prior to calculating the below medians and IQRs. There was one additional patient in the thiamine group whose lactate at 48-hours was not imputed as it was missing due to non-death reasons, leading to n = 17 for thiamine (instead of 18).
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | Thiamine | Placebo
Number analyzed (Participants) | 17 | 18
mmol/L | 1.9 [1.1 to 7.5] | 1.8 [1.2 to 5.4]
Statistical Analysis 1: Comparison: Thiamine vs Placebo; Test type: Other — Linear mixed-effects model with an independent variance-covariance matrix to account for the correlation of within-patient repeated measures was used and linear contrasts were used to estimate the mean difference between treatment arms at 48 hours; p = 0.9, Mixed Models Analysis — Global p-value from the mixed model; If patients died before 48 hours lactate levels were imputed by carrying forward the last known value before the event with a 20% increase; Mean Difference (Final Values) = 1.5, 95% CI 2-sided [-3.1 to 6.1]

2. Secondary Outcome: Oxygen Consumption
Description: The investigators will evaluate the mean oxygen consumption over two days, compared between groups
Time Frame: 2 days
Population: 22 patients had metabolic data at 48 hours, n = 11 in placebo, n = 11 in thiamine
Measure: Mean (Standard Deviation); unit: Area under the Curve VO2 (mL/kg/min)
Arm/Group | Thiamine | Placebo
Number analyzed (Participants) | 11 | 11
Area under the Curve VO2 (mL/kg/min) | 3.83 (0.94) | 3.48 (1.27)
Statistical Analysis 1: Comparison: Thiamine vs Placebo; AUC-VO2 normally distributed, used a linear regression model to compare mean AUC-VO2 between treatment groups controlling for average temperature; Test type: Other; p = 0.42, Regression, Linear; Mean Difference (Final Values) = -0.36, 95% CI 2-sided [-1.29 to 0.56]

3. Secondary Outcome: Pyruvate Dehydrogenase
Description: The investigators will evaluate the median pyruvate dehydrogenase levels over two days, compared between groups
Time Frame: 2 days
Population: Only 12 patients in Thiamine and 13 patients in Placebo alive and with non-missing PDH specific activity values at 48-hours.
Measure: Median (Inter-Quartile Range); unit: mini OD unit/min/mg protein
Arm/Group | Thiamine | Placebo
Number analyzed (Participants) | 12 | 13
mini OD unit/min/mg protein | 1.2 [0.9 to 1.5] | 1.1 [1.0 to 1.3]
Statistical Analysis 1: Comparison: Thiamine vs Placebo; Test type: Other; p = 0.07, Mixed Models Analysis — Mixed model controlling for repeated measures within patients used to get a mean difference in PDH specific activity between thiamine and placebo groups at 48 hours; P-value is the global p-value from the mixed model; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.9 to 0.3]

ADVERSE EVENTS:
Time Frame: From enrollment to time of hospital discharge or 90 days, whichever is first.
Arm/Group | Thiamine | Placebo
All-Cause Mortality (participants affected / at risk) | 12/18 | 12/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

LIMITATIONS AND CAVEATS:
The trial was placed on hold after a data safety and monitoring board (DSMB) review noted possible harm from thiamine in the subgroup of patients with a lactate >5mmol/L at the time of study inclusion, with a similar pattern seen in a companion trial in out-of-hospital cardiac arrest (NCT03450707). While the option of continuing to enroll patients with lactate ≤ 5mmol/L was provided, the trial was terminated formally in August 2022 due to lack of feasibility.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-04): https://cdn.clinicaltrials.gov/large-docs/57/NCT02974257/Prot_SAP_000.pdf